CLINICAL TRIAL: NCT00550901
Title: Phase I Study of Cis-Diamminedicholoroplatinum in Combination With ICRF-187 in the Treatment of Advanced Malignancies
Brief Title: Dexrazoxane and Cisplatin in Treating Patients With Advanced Solid Tumors
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: City of Hope Medical Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Stephen Shibata M.D. Principal Investigator, City of Hope Medical Center
Purpose: Treatment
Other Study IDs: CDR0000570420; P30CA033572 (NIH); CHNMC-00136
Record Dates: First submitted 2007-10-25; First posted 2007-10-30 (Estimated); Last update posted 2015-06-08 (Estimated); Status verified 2015-06

CONDITIONS: Unspecified Adult Solid Tumor, Protocol Specific
Keywords: unspecified adult solid tumor, protocol specific
MeSH Terms: interventions — Cisplatin; Dexrazoxane; Chromatography, High Pressure Liquid; Mass Spectrometry

INTERVENTIONS:
Drug: cisplatin
Drug: dexrazoxane hydrochloride
Other: high performance liquid chromatography
Other: laboratory biomarker analysis
Other: mass spectrometry
Other: pharmacological study

SUMMARY:
RATIONALE: Drugs used in chemotherapy, such as dexrazoxane and cisplatin, work in different ways to stop the growth of tumor cells, either by killing the cells or by stopping them from dividing. Giving more than one drug (combination chemotherapy) may help kill more tumor cells.

PURPOSE: This phase I trial is studying the side effects and best dose of dexrazoxane when given together with cisplatin in treating patients with advanced solid tumors.

DETAILED DESCRIPTION:
OBJECTIVES:

* To establish the maximum tolerated dose of a 96-hour continuous infusion of dexrazoxane hydrochloride and a single-dose, one-hour infusion of cisplatin in patients with advanced solid tumors.
* To determine the pharmacokinetics of dexrazoxane hydrochloride and cisplatin when given concurrently.
* To describe the toxicities of infusional dexrazoxane hydrochloride and cisplatin given in combination.

OUTLINE: Patients receive dexrazoxane hydrochloride IV continuously over 96 hours beginning on day 1 and cisplatin IV over 1 hour on day 3. Courses repeat every 21 days in the absence of disease progression or unacceptable toxicity.

Blood is collected periodically during course one for pharmacokinetic studies. DNA isolated from the samples is also analyzed for oxidative DNA damage by gas chromatography/mass spectrometry.

After completion of study treatment, patients are followed periodically.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

Inclusion criteria:

* Histologically confirmed advanced, incurable cancer that is unresponsive to prior chemotherapy regimens or for which no standard chemotherapy regimen exists
* History of brain metastases allowed if controlled by radiotherapy or surgery and patient's neurological status is stable

  * Concurrent corticosteroids allowed as long as required dose is stable or decreasing
* Not eligible for a higher priority study

PATIENT CHARACTERISTICS:

Inclusion criteria:

* Karnofsky performance status 60-100%
* Life expectancy ≥ 12 weeks
* ANC ≥ 2,000/mm³
* Platelet count ≥ 100,000/mm³
* Serum creatinine ≤ 1.6 mg/dL OR creatinine clearance ≥ 60 mL/min
* Bilirubin ≤ 1.5 mg/dL
* SGOT < 3 times upper limit of normal
* Recovered from any recent severe infection
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception

Exclusion criteria:

* Patients with any nonmalignant intercurrent illnesses (e.g., cardiovascular, pulmonary, neurologic) that are either poorly controlled with currently available treatment, or are of such severity that the investigators deem it unwise to enter the patient onto this study

PRIOR CONCURRENT THERAPY:

Inclusion criteria:

* See Disease Characteristics
* At least 4 weeks since prior radiotherapy or chemotherapy and recovered
* Recovered from prior major surgery

Exclusion criteria:

* Concurrent treatment for severe infection

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Estimated)
Dates: Start 2001-02; Primary Completion 2007-07 (Actual); Study Completion 2007-07 (Actual)

PRIMARY OUTCOMES:
Toxicity
Maximum tolerated dose of dexrazoxane hydrochloride and cisplatin

CONTACTS AND LOCATIONS:
Overall Officials: Stephen I. Shibata, MD, Study Chair — City of Hope Comprehensive Cancer Center